CLINICAL TRIAL: NCT05639569
Title: Ankura™ TAA Stent Graft System Post-Market Clinical Follow-up Study: Multi-center, Prospective, Observational, Post-Market Follow-up Study
Brief Title: Ankura™ TAA Stent Graft System Post-Market Clinical Follow-up Study
Status: Recruiting | Type: Observational
Sponsor: Lifetech Scientific (Shenzhen) Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: LT/TS/12C-2021-01
Record Dates: First submitted 2022-11-26; First posted 2022-12-06 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Aneurysm Thoracic; Dissection of Thoracic Aorta
MeSH Terms: conditions — Aortic Aneurysm, Thoracic; Dissection, Thoracic Aorta

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Descending Thoracic Aneurysm (DTA) or Type B Aortic Dissection (TBAD): All patients who signed informed consent and are used with Ankura™ TAA Stent Graft Systems will undergo follow-up (FU) evaluations as per local hospital standards and corresponding IFU which is expected to be at the following time points post-implant:
  Before discharge, 30days after the procudure, 3-6 months after the Procedure, 12 months after the procedure, 24 months after the procedure, 36 months after the procedure
  Interventions: Device: Ankura™ TAA Stent Graft System

INTERVENTIONS:
Device: Ankura™ TAA Stent Graft System — All patients will be implanted with Ankura™ TAA Stent Graft System in accordance with the instructions for use (IFU).

SUMMARY:
The purpose of this study is to collect clinical data on patient outcomes, evaluate the safety and performance of Ankura TAA Stent Graft System and Surpass Super Stiff Guidewire, and build clinical evidence for patients with Descending Thoracic Aneurysm (DTA) or Type B Aortic Dissection (TBAD).

DETAILED DESCRIPTION:
The physician shall strictly follow the clinical study protocol and shall not deviate from or substantially change the protocol. However, in case of emergency such as immediate risk to the subjects, which needs tobe eliminated immediately, it may be reported in written form afterwards. During the course of the study,documents such as amendments to the clinical study protocol and informed consent, requests for deviation,and resumption of the suspended clinical study shall be subject to the written approval of the Ethics Committee

ELIGIBILITY:
Inclusion Criteria:

* Patient has descending thoracic aortic aneurysm (DTA) or type B aortic dissection (TBAD), who needs endovascular repair (TEVAR).
* Life expectancy > 1 year.
* Patient or legally authorized representative understands the nature of the clinical trial, agrees to its provisions, agrees to comply with the requirements of the study including a 3-year follow-up, and signed applicable Informed Consent Form.
* Patient's characteristics consistent with Ankura™ Stent Graft System IFU and sizing guidelines, which indicate as following:

  1. For descending thoracic aortic aneurysm (DTA) patient:

     * Adequate iliac/femoral access vessel that is compatible with the required delivery system.
     * Aortic inner diameter in the range of 18-42mm.
     * ≥15mm non-aneurysmal aorta proximal and distal to the lesion.
     * Morphology suitable for endovascular repair.
  2. For type B aortic dissection (TBAD) patient:

     * Adequate iliac/femoral access vessel that is compatible with the required delivery system.
     * ≥15mm landing zone proximal to the primary entry tear; proximal extent of the landing zone must not be dissected. Diameter at proximal extent of proximal landing zone in the range of 16-44mm.
     * ≥15mm landing zone distal to the primary entry tear; distal extent of the landing zone must not be dissected. Diameter at distal extent of distal landing zone in the range of 16-44mm.
     * Morphology suitable for endovascular repair.

Exclusion Criteria:

* Patient with any contraindications mentioned in the Ankura™ Stent Graft System IFU:

  * Patients with acute systemic infection;
  * Patients who have had other devices implanted in the cardiovascular cavity, which will interfere with the placement of this device;
  * Patients with mesenteric blood flow mainly supplied by the inferior mesenteric artery;
  * Patients who have allergic reaction to the device;
  * Patients who are not suitable for endovascular repair in vascular morphology;
  * Patients who cannot tolerate contrast agents due to severe renal insufficiency;
  * Patients who are allergic to contrast agents;
  * Aneurysms neck with thrombus;
  * Non-aneurysmal aortic proximal neck length <1.5cm;
  * Non-aneurysmal aortic distal anchorage zone <1.5cm;
  * For aneurysms, Non-aneurysmal aortic diameter <18mm or >42mm. For Type B dissections, Non-aneurysmal aortic diameter <16mm or >44mm.
* Patient with traumatic aortic injury;
* Patient with uncorrectable coagulopathy;
* Patient with hereditary connective tissue disease, including but not limited to Marfan Syndrome or Ehlers-Danlos Syndrome;
* Patient with morbid obesity, weight greater than 350 Pounds (150kg), or who cannot undergo accurate fluoroscopy examination due to obesity;
* Age<18 Years or Age> 85 Years;
* Pregnant or plan to be pregnant or breast feeding;
* Myocardial infarction or stroke within 3 months prior to the procedure;
* American Society of Anesthesiologists Physical Status Classification (ASA) classification 5 or higher;
* Patient with an unstable angina pectoris or hearth insufficiency New York Heart Association Functional Classification (NYHA) 3 or 4
* Participant in other drug or medical device clinical trials;
* Patient with access vessel which are to tortuous, narrow or any kind of reasons that would lead to failure of introduction and advancing an introducer sheath;
* Any condition (medical or anatomic) which makes the patient not suitable for endovascular repair according to the opinion of the investigator.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Descending Thoracic Aneurysm (DTA) or Type B Aortic Dissection (TBAD) and indicate for endovascular repair (TEVAR).
Sampling Method: Non-Probability Sample
Enrollment: 145 (Estimated)
Dates: Start 2023-05-03 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of major adverse events | Timeframe: within 30-day post-implantation
  Incidence of major adverse events.
Freedom from stent graft-related events | Timeframe: within 12-month post-implantation
  Freedom from stent graft-related events (12 months)

CONTACTS AND LOCATIONS:
Locations (8):
- Germany (3):
  - RHÖN-KLINIKUM Campus Bad Neustadt, Bad Neustadt an der Saale
  - Asklepios Klinik Nord Heidberg, Hamburg
  - St. Franziskus Hospital Münster, Münster
- Greece (3):
  - Evaggelismos General Hospital, Athens
  - General Hospital of Athens - Georgios Gennimatas, Athens
  - University General Hospital - Attikon, Attiki
- A.O. Ordine Mauriziano di Torino, Turin, Italy
- Federal State Budgetary Institution - V.A. Almazov National Medical Research Centre, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No